CLINICAL TRIAL: NCT06602297
Title: A Prospective, Single-center, Cross-sectional Clinical Investigation of Propofol-related Euphoria in Pain-free Gastrointestinal Endoscopy Patients
Brief Title: Propofol-related Euphoria in Pain-free Gastrointestinal Endoscopy Patients
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Study Director, Northern Jiangsu People's Hospital
Other Study IDs: 2024ky248
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Propofol; Addictive Behaviors
MeSH Terms: conditions — Behavior, Addictive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To define the prevalence, duration and severity of propofol-associated euphoria in patients undergoing painless gastrointestinal endoscopy and to explore the independent influencing factors by means of a single-center, cross-sectional clinical research study

ELIGIBILITY:
Inclusion Criteria:

* Proposed to perform painless GI endoscopy, and simple endoscopic maneuvers such as single small polyp clamping, performing HP examination, etc;
* Gender is not limited;
* 18 years old ≤ 80 years old;
* ASA classification: I-II;
* 18 kg/m2 <BMI <30 kg/m2;
* Informed consent, voluntary participation in the trial, and informed consent signed by the subjects themselves.

Exclusion Criteria:

* adjudicated respiratory management difficulties;
* History of substance abuse as well as drug use;
* Participation in a clinical trial of another drug or device within 3 months prior to the screening period
* Use of therapeutic drugs (e.g., benzodiazepines, opioid analgesics) by the subject within 3 months prior to the Screening Period for a variety of reasons (e.g., insomnia, pain, etc.) that may have an impact on the outcome of the trial, etc;
* Allergy or contraindication to the study drug or components thereof;
* Previous psychiatric or neurological disorders (e.g., schizophrenia, mania, bipolar disorder, psychosis, epilepsy, neuralgia, etc.) and a history of taking medications corresponding to the treatment of the corresponding psychiatric or neurological disorders (e.g., antidepressants, anxiolytics, convulsants, antiepileptic drugs, etc.);
* Pregnant women;
* Subjects with severe communication disorders due to severe hearing deterioration;
* Refusal to participate in this study;
* Those deemed unsuitable by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Participants with ASA I-II Proposed for Painless Gastrointestinal Endoscopy
Sampling Method: Probability Sample
Enrollment: 986 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of propofol-related euphoria | preoperatively , within half an hour after the operation, postoperative days 1 ,3 and 7
  Subjects were asked in person or through telephone follow-up, "To what extent do you think you are feeling pleasure and euphoria now?". The NRS is a numerical rating scale (NRS) that represents feelings of euphoria on a scale of 0-10, with 0 being no feelings of euphoria at all and 10 being the strongest feelings of euphoria.
Severity of propofol-related euphoria | preoperatively , within half an hour after the operation, postoperative days 1,3 and 7
  Subjects were asked in person or via telephone follow-up, "Has your pleasant, euphoric mood changed now compared to before surgery?" , using the Likert questionnaire score (5-Point Likert Scale, Likert): 0 indicates that the mood is significantly worse than before; 1 indicates that the mood is mildly worse than before; 2 indicates that there is no change in euphoria; 3 indicates that there is a mild euphoria; and 4 indicates that there is a markedly euphoric mood.
Duration of propofol-related euphoria | within half an hour after the operation, postoperative days 1 ,3 and 7
  Postoperatively, subjects were asked about changes in mood compared to baseline values by the same method, and their duration was confirmed.

SECONDARY OUTCOMES:
Anxiety level | preoperatively , within half an hour after the operation, postoperative days 1,3 and 7
  Face-to-face questioning or follow-up via telephone, questioning the disease to record the anxiety level, using the NRS rating, which represents the anxiety level through ten numbers from 0-10, with 0 being no anxiety at all and 10 being the most intense anxiety.
Subject satisfaction with the quality of perioperative anesthesia | at postoperative days 1 after the subject had recovered from all adverse events, if the subject did not have a perioperative adverse event
  Assessment method: in person or through telephone follow-up, the subjects were asked to measure their satisfaction with the intraoperative and postoperative resuscitation periods as well as the entire period after discharge, which was rated by NRS, and satisfaction was represented by ten numbers from 0-10, with 0 being unsatisfactory and 10 being the most satisfactory.
Content of Memory of Intraoperative Dreams | Within half an hour after the operation
  If the subject was able to recall the dream, the dream was rated on a Likert questionnaire: 1. the mood of the dream: 1-5, 1 as very sad, 5 as very happy; 2. the extent to which the dream was remembered; 1-5, 1 as not remembering at all, 5 as remembering at all: 3. the sounds in the dream: 1-5, 1 as not at all, 5 as all of them; 4. the movements in the dream: 1-5 1 for not at all, 5 for all of them.
  Calculate the sum of the Dreamland Likert questionnaire scores.
The number of times of sleep in the 72h postoperative period | Postoperative days 1 and 3
  The number of times of sleep were asked and recorded during the 72h period after painless gastrointestinal endoscopy by telephone follow-up.
the duration of each sleep in the 72h postoperative period | Postoperative days 1 and 3
  The duration of each sleep were asked and recorded during the 72h period after painless gastrointestinal endoscopy by telephone follow-up.
the quality of sleep each time in the 72h postoperative period | Postoperative days 1 and 3
  Ask for and record the quality of sleep each time through telephone follow-ups The quality of sleep was categorized into five grades of "very good, good, fair, bad, and very bad" . Each grade corresponds to 5, 4, 3, 2, and 1 points.
Perioperative adverse events | Within half an hour after the operation, postoperative days 1,3 and 7. If the adverse events had not disappeared by T7d, telephone follow-up was conducted every 3d thereafter until the adverse events were resolved.
  In-person questioning or telephone follow-up, using the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, to determine perioperative adverse events and assess the severity of the adverse events against the feedback collected from the subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China